CLINICAL TRIAL: NCT01976715
Title: Characterization and Management of Patients With HIV-1 Infection Who Experience Virologic Failure Despite Combination Antiretroviral Therapy
Brief Title: Study of People With HIV Infection Who Have High Viral Loads Despite Combination Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140009; 14-I-0009
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Acquired Immune Deficiency Syndrome Virus; Acquired Immunodeficiency Syndrome Virus; AIDS Virus; Human Immunodeficiency Virus; Human Immunodeficiency Viruses
Keywords: HIV; Treatment Failure; Drug Resistance; Natural History
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-1: Subjects (greater than or equal to 18 years) with human immunodeficiency virus type 1 (HIV-1) who have documented virologic failure.

SUMMARY:
Background:

- The human immunodeficiency virus (HIV) causes acquired immune deficiency syndrome (AIDS). Combination antiretroviral therapy (ART) drugs treat HIV infection. They generally decrease the amount of HIV virus in the blood (called viral load) to very low levels. This happens only if the drugs still fight HIV and if taken every day exactly as prescribed. When not taken as directed, or if the ART drugs are not strong enough, the virus can become resistant to them, and the ART will not work to control the virus. Researchers want to know how to control HIV in people who can t lower their viral load with their current ART drugs.

Objective:

-<TAB>To better control HIV in people who can t get a lower viral load even with ART drugs and to learn more about why the HIV is not under control.

Eligibility:

* People at least 18 years old and with HIV.
* People who have been on at least two combinations of ART drugs (including current ART).
* People whose last two viral loads were greater than 1,000 copies/mL.

Design:

* Participants will be screened with medical history, physical exam, and blood tests.
* Participants will then have a baseline visit. They will have another physical exam, blood tests, plus answer questions about what they know about HIV and ART, and how they take their ART.
* Participants will arrange to stay in the NIH hospital for 7 8 days.
* They will take their medications as usual. At the time to take the ART drugs, they will have to ask a nurse to bring them. If they forget, the nurse will bring them.
* Participants will meet with a doctor, pharmacist, social worker and nurse to discuss ways to help participants remember to take their drugs.
* Participants will have blood drawn about every other day.
* Researchers will study the test results. Some participants will be put on different ART drugs. If that happens, participants will have another NIH hospital stay for 7-8 days.
* Participants will have 4 follow-up visits over 12 weeks, then every 3 months for 2 years or more.

DETAILED DESCRIPTION:
Combination antiretroviral therapy (ART) has dramatically improved survival in individuals with human immunodeficiency virus type1 (HIV-1) infection. Despite recent development of more potent regimens with fewer toxicities and lower pill burden, there remains a subpopulation of subjects who fail to achieve and maintain viral suppression while on treatment. Factors known to contribute to virologic failure include suboptimal adherence, drug resistance, suboptimal regimen potency, sequential introduction of single drugs to a failing regimen, and reduced ART exposure due to impaired drug absorption or pharmacokinetic drug-drug interactions.

This is a natural history protocol with intensive observation intended to characterize and manage HIV-infected subjects who have documented virologic failure on their current regimen and who have experienced virologic failure in meeting one of the following criteria:

1. Documented virologic failure on at least 1 prior ART regimen and at least 2 consecutive HIV RNA plasma measurements of >1,000 copies/mL, including the last documented value, while on the current prescribed ART regimen for at least 6 months; or
2. Documented extensive resistance to at least 3 ARV drug classes, and has persistent plasma viremia (HIV RNA > 1,000 copies/mL for > 6 months) despite multiple regimen changes, regardless of how long the subject has been prescribed his or her current regimen.

We anticipate that, for a large proportion of the participants enrolled in this protocol, non-adherence, with or without drug resistance, is the most common reason for the virologic failure. Another objective for the study is to assess the impact of a 7-day, self-guided, inpatient directly observed therapy (iDOT) or a 7-day outpatient, self-guided electronic directly observed therapy (eDOT) on HIV RNA kinetics, when participants will receive their pre-enrollment ART regimens. During the iDOT period, participants will request their ARV drugs at a pre-arranged time reflecting their home medication schedule. Failure to do so will be recorded and the medications will then be provided by the nursing staff. Blood draw will be done on days 1, 3, 5, and 8. Participants will be discharged on Day 8 after morning blood draw. During the eDOT period, participants will submit video recordings of themselves taking their medications at the scheduled time for 7 days. Reminders (eg, short message service [SMS], push notifications) will be sent to participants if they have not submitted their video recordings 2 hours past the scheduled time . Participants who use eDOT will present to the NIH Clinical Center on Day 1 and return on Day 8 to have blood draw for HIV RNA and safety labs as per protocol. Adherence and psychosocial assessments will also be performed. Plasma concentrations from at least one of the ARV drugs in the regimen will be measured on the first and last day of iDOT/eDOT to determine if suboptimal drug plasma concentration was a contributing factor to virologic failure.

Within approximately 2 weeks, but no later than 4 weeks, after iDOT/eDOT (post-iDOT/eDOT phase), the research team will review the results from the HIV-1 viral load kinetics, current and cumulative genotypic and/or phenotypic resistance tests, ART history and responses, and other identified factors that could have contributed to the treatment failure (such as concomitant medications, history of antiretroviral adverse events, and psychosocial barriers). The team will then design a new, individualized treatment plan for each participant. Participants will either continue on their pre-enrollment ART regimen, or they will receive a new, individually tailored regimen that consists of FDA-approved ARVs.

Alternatively, participants may co-enroll on a clinical trial for investigational ARVs, or may receive expanded access treatment, if either option is available.

New regimens initiated due to virologic failure will be monitored during a subsequent 7-day, self-guided iDOT or 7-day self-guided eDOT. Participants will be followed after the iDOT/eDOT at weeks 2 (plus/minus 3 working days), 4 (plus/minus 3 working days), 8 (plus/minus 7 days), and 12 (plus/minus 7 days), and then every 3 months (plus/minus 2 weeks) for up to 2 years, with the option of extending participation longer if there is continued research interest as identified by the study team. The same treatment plan may be repeated if a participant fails to respond to a new regimen.

In a select group of subjects who fail to achieve viral suppression, advanced HIV-1 variant analysis may be used to attempt to identify the presence of minority drug resistant variants. This analysis will be used as supplemental information to construct new regimens for this group of participants. Samples of plasma, serum, and peripheral blood mononuclear cells will be stored for further evaluation of virologic evolution and other factors that may be contributing to treatment failure in this population.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age, greater than or equal to 18 years.
  2. Documented HIV-1 infection (prior written documentation such as positive standard ELISA or rapid HIV-1/HIV-2 antibody test with confirmatory Western Blot, or documentation of repeated HIV RNA of greater than 1,000 copies/mL)..
  3. Established care with an HIV primary care provider.
  4. Fulfilling one of the following criteria for virologic failure:

     1. Documented virologic failure on at least 1 prior ART regimen and at least 2 consecutive HIV RNA plasma measurements of greater than 1,000 copies/mL, including the last documented value, while on the current prescribed ART regimen for at least 6

        months; or
     2. Documented extensive resistance to at least 3 ARV drug classes, and has persistent plasma viremia (HIV RNA greater than 1,000 copies/mL for greater than 6 months) despite multiple regimen changes, regardless of how long the subject has been prescribed his or her current regimen.
  5. Willingness to have samples stored for future research.
  6. Willingness to undergo genetic testing.
  7. Ability and willingness to provide informed consent
  8. Willingness to be hospitalized for iDOT or record videos of themselves for eDOT.

EXCLUSION CRITERIA:

1. HIV RNA levels at screening <1,000 copies/mL.
2. Receiving medical care for an acute medical illness stemming from a significant comorbidity; enrollment may be deferred or postponed until the condition resolves or stabilizes.
3. Pregnancy (if a subject becomes pregnant while enrolled in the protocol, she will continue participation throughout her pregnancy).
4. Any illness or condition that, in the investigator s opinion, may substantially increase the risk associated with the subject s participation in the study, or may compromise the scientific objectives.

NOTE: Participants will not be excluded based on stable laboratory abnormalities, hepatitis B virus (HBV) or hepatitis C virus (HCV) co-infection status, etc. Selection of a new ART regimen will account for any co-existing conditions, such as known risks of antiretroviral drugs to the fetus, dosage adjustment due to organ dysfunction, drug interaction potential with concomitant agents, and the need for treatment of HBV co-infection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
The log viral load change over time during the study enrollment period | 2 years after enrollment
  viral load

SECONDARY OUTCOMES:
Log viral load change during the inpatient directly observed therapy period | After DOT hospitalization
  viral load

CONTACTS AND LOCATIONS:
Overall Officials: Alice K Pau, Pharm.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ortiz R, Dejesus E, Khanlou H, Voronin E, van Lunzen J, Andrade-Villanueva J, Fourie J, De Meyer S, De Pauw M, Lefebvre E, Vangeneugden T, Spinosa-Guzman S. Efficacy and safety of once-daily darunavir/ritonavir versus lopinavir/ritonavir in treatment-naive HIV-1-infected patients at week 48. AIDS. 2008 Jul 31;22(12):1389-97. doi: 10.1097/QAD.0b013e32830285fb. PMID 18614861
- [Background] Harrison KM, Song R, Zhang X. Life expectancy after HIV diagnosis based on national HIV surveillance data from 25 states, United States. J Acquir Immune Defic Syndr. 2010 Jan;53(1):124-30. doi: 10.1097/QAI.0b013e3181b563e7. PMID 19730109
- [Background] Johnson LF, Mossong J, Dorrington RE, Schomaker M, Hoffmann CJ, Keiser O, Fox MP, Wood R, Prozesky H, Giddy J, Garone DB, Cornell M, Egger M, Boulle A; International Epidemiologic Databases to Evaluate AIDS Southern Africa Collaboration. Life expectancies of South African adults starting antiretroviral treatment: collaborative analysis of cohort studies. PLoS Med. 2013;10(4):e1001418. doi: 10.1371/journal.pmed.1001418. Epub 2013 Apr 9. PMID 23585736
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-I-0009.html